CLINICAL TRIAL: NCT02321150
Title: A Novel Technique for the Removal of Pterygiums
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Dr. Kim Jebodhsingh, Consultant Ophthalmologist, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KJebodhsingh
Record Dates: First submitted 2014-12-03; First posted 2014-12-22 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Pterygium
Keywords: Pterygium; Pterygiums; Pterygia; Graft; Autograft; Excision; Surgery; Eye; electrocautery; polyglactin
MeSH Terms: conditions — Pterygium | interventions — Cautery; Sutures; Polyglactin 910

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sutures (Active Comparator): After pterygium removal the conjunctival graft to cover bare sclera will be secured with interrupted 8.0 polyglactin sutures.
  Interventions: Procedure: Sutures
- Cautery (Experimental): After pterygium removal the conjunctival graft to cover bare sclera will be secured with bipolar electrocautery, power set at 25 until whitening of tissue observed.
  Interventions: Procedure: Cautery

INTERVENTIONS:
Procedure: Cautery — * Pterygium dissected off, corneal bed burred smooth and autograft harvested as per usual technique.
  * Conjunctiva undermined at the recipient site.
  * Relaxing incisions placed at the corners of the recipient site.
  * Graft is slid into place
  * Graft / host interface is gently dried with a Qtip
  * Bipolar cautery is applied after grasping the graft and host conjunctiva gently between cautery forceps.
    * Power setting: 25.
    * Duration of cautery: 4 -5 seconds; the tissue should whiten and contract as desiccation and coagulation take place. Some charring may occur.
  * Counter traction is applied to the conjunctiva as the cautery forceps are gently teased off
  * Cautery is applied at the 4 apices of the graft then in between these points.
  Other Names: Mentor O&O Wetfield Coagulator
  Arms: Cautery
Procedure: Sutures — * Pterygium dissected off, corneal bed burred smooth and autograft harvested as per usual technique.
  * Conjunctiva undermined at the recipient site.
  * Graft is slid into place The graft is secured to host conjunctiva using 7 interrupted sutures
  Other Names: Polyglactin, Vicryl
  Arms: Sutures

SUMMARY:
The aim of this study is to introduce a new surgical technique for the removal of pterygiums that entails the use of bipolar electrocautery to secure the graft, rather than sutures.

With this, the objective is to evaluate the benefits of a new technique for pterygium surgery with respect to postoperative patient comfort, surgery time, cost and recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more pterygiums over age 18

Exclusion Criteria:

* Patients with glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Patient Discomfort | Day 1
  Grading of patients' symptoms (pain, foreign body sensation, irritation, and epiphora) will be done using a 5-point scale. The scale ranges from 0 to 4:
  0 = no symptom at all;
  1. = presence of the symptom but easily tolerated;
  2. = presence of the symptom causing some discomfort;
  3. = presence of the symptom causing discomfort that interferes with usual activity or sleep;
  4. = presence of the symptom that completely interferes with usual activity or sleep.
Patient Discomfort | Week 1
  Grading of patients' symptoms (pain, foreign body sensation, irritation, and epiphora) will be done using a 5-point scale. The scale ranges from 0 to 4:
  0 = no symptom at all;
  1. = presence of the symptom but easily tolerated;
  2. = presence of the symptom causing some discomfort;
  3. = presence of the symptom causing discomfort that interferes with usual activity or sleep;
  4. = presence of the symptom that completely interferes with usual activity or sleep.
Patient Discomfort | Week 2
  Grading of patients' symptoms (pain, foreign body sensation, irritation, and epiphora) will be done using a 5-point scale. The scale ranges from 0 to 4:
  0 = no symptom at all;
  1. = presence of the symptom but easily tolerated;
  2. = presence of the symptom causing some discomfort;
  3. = presence of the symptom causing discomfort that interferes with usual activity or sleep;
  4. = presence of the symptom that completely interferes with usual activity or sleep.
Patient Discomfort | Week 3
  Grading of patients' symptoms (pain, foreign body sensation, irritation, and epiphora) will be done using a 5-point scale. The scale ranges from 0 to 4:
  0 = no symptom at all;
  1. = presence of the symptom but easily tolerated;
  2. = presence of the symptom causing some discomfort;
  3. = presence of the symptom causing discomfort that interferes with usual activity or sleep;
  4. = presence of the symptom that completely interferes with usual activity or sleep.
Patient Discomfort | Week 7
  Grading of patients' symptoms (pain, foreign body sensation, irritation, and epiphora) will be done using a 5-point scale. The scale ranges from 0 to 4:
  0 = no symptom at all;
  1. = presence of the symptom but easily tolerated;
  2. = presence of the symptom causing some discomfort;
  3. = presence of the symptom causing discomfort that interferes with usual activity or sleep;
  4. = presence of the symptom that completely interferes with usual activity or sleep.
Patient Discomfort | 3 months
  Grading of patients' symptoms (pain, foreign body sensation, irritation, and epiphora) will be done using a 5-point scale. The scale ranges from 0 to 4:
  0 = no symptom at all;
  1. = presence of the symptom but easily tolerated;
  2. = presence of the symptom causing some discomfort;
  3. = presence of the symptom causing discomfort that interferes with usual activity or sleep;
  4. = presence of the symptom that completely interferes with usual activity or sleep.

SECONDARY OUTCOMES:
Operating time | day 1
  Analysis. start time of operation, start time of conjunctival graft attachment and end time of operation will be recorded.

OTHER OUTCOMES:
Operating Cost | day 1
  Cost Benefit Analysis. Total cost of pterygium surgery using sutures for graft attachment versus cost using cautery for graft attachment will be calculated and compared.
Recurrence | 1 year
  Any regrowth of the pterygium onto the cornea will be considered a recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Kim N Jebodhsingh, MBBS, DABO, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Bridgetown, Barbados